CLINICAL TRIAL: NCT06288841
Title: Efficacy and Safety of Liposomal Bupivacaine Under ERAS Concept for Postoperative Analgesia of Ultrasound-Guided QLB in Gynecologic Laparoscopic Patients: A Randomized, Single-blind, Active-Controlled Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Ning Luo, Resident Doctor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJMZ2023-008
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Pharmacological Action
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ropivacaine injection group (Placebo Comparator)
  Interventions: Drug: Ropivacaine injection
- Bupivacaine liposomal low-dose group (Experimental)
  Interventions: Drug: Bupivacaine liposome
- Bupivacaine liposomal medium-dose group (Experimental)
  Interventions: Drug: Bupivacaine liposome
- Bupivacaine liposomal high-dose group (Experimental)
  Interventions: Drug: Bupivacaine liposome

INTERVENTIONS:
Drug: Ropivacaine injection — Ultrasound-guided bilateral QLB2 was performed using Ropivacaine injection prior to anesthesia induction
  Other Names: Quadratus lumborum block
  Arms: Ropivacaine injection group
Drug: Bupivacaine liposome — Ultrasound-guided bilateral QLB2 was performed using Bupivacaine liposome injection prior to anesthesia induction
  Other Names: Quadratus lumborum block
  Arms: Bupivacaine liposomal high-dose group; Bupivacaine liposomal low-dose group; Bupivacaine liposomal medium-dose group

SUMMARY:
With the development of the concept of comfortable medicine and enhanced recovery surgery (ERAS), optimizing the perioperative management of patients, reducing surgical stress, and reducing postoperative pain can effectively reduce perioperative complications and achieve the purpose of accelerating recovery. As an important part of ERAS, multimodal analgesia is the core concept of perioperative analgesia management. As a kind of perioperative multimodal analgesia, quadratus lumbar muscle block (QLB) is a type of local anesthetic drug injected around the quadratus lumbar muscle to reduce or eliminate abdominal wall pain and visceral pain after abdominal surgery. QLB has been used successfully for pain control after laparoscopic and open surgery, reducing perioperative opioid use and improving prognosis-related measures such as PONV and length of hospital stay. Bupivacaine liposomes use DepoFoam technology to encapsulate the drug in polycystic liposomes, which can prolong the release time of bupivacaine due to the different rupture times of different vesicles, and the postoperative analgesia can be up to 72 hours. In this project, patients who undergo elective laparoscopic uterine and double adnexectomy were selected to be injected with lipososomes of bupivacaine at different concentrations under ultrasound guidance of bilateral posterior QLB before anesthesia induction, and the effect of liposomal bupivacaine on postoperative pain was investigated by evaluating the postoperative pain and incidence of adverse events. This study will greatly promote the clinical promotion and application of bupivacaine liposome, improve the postoperative comfort and satisfaction of patients, and accelerate the postoperative recovery of patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-65 years; 2) ASA grade I or II; 3) Patients who are scheduled to undergo elective laparoscopic hysterectomy or laparoscopic hysterectomy and double adnexectomy; 4) BMI of 19-29 kg/m2; 5) Patients who voluntarily sign the informed consent form.

Exclusion Criteria:

* 1) Those who are known to be allergic to the drug components of this study and have allergic constitution; 2) History of allergy to general anesthetic drugs, opioids, and non-steroidal drugs; 3) Patients who need to switch to laparotomy for various reasons; 4) history of neurological disease; History of chronic pain; drug addiction and alcohol abuse; History of long-term opioid use; Opioids are given 48 hours before surgery; 5) ASA grade III or IV; 6) Coronary heart disease, bronchial asthma, severe hypertension, severe hematologic dysfunction, liver and kidney function, and obvious abnormalities in electrolytes; 7) Patients with severe gastrointestinal diseases; 8) Patients who refuse to use intravenous PCIA for analgesia; 9) Pregnant or lactating women; 10) Patients with infection in the skin of the abdominal injection area; 11) Patients with rheumatoid or inflammatory arthritis or diseases requiring chronic analgesic treatment; 12) Patients who have been treated for deep vein thrombosis, pulmonary embolism, myocardial infarction or ischemic stroke in the past 6 months; 13) Those who have poor compliance and cannot complete the test according to the research protocol; 14) Those who have participated in clinical trials of other drugs in the past 4 weeks; 15) Any circumstances that, in the opinion of the investigators, are not suitable for inclusion.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-11-29 (Estimated)

PRIMARY OUTCOMES:
NRS pain score within 72 hours after surgery | Postoperative (starting from the end of the operation) 2 hours (h), 4h, 6h, 8h, 12h, 24h, 48h, 72h
  After surgery (starting from the end of surgery), NRS was evaluated at 2h, 4h, 6h, 8h, 12h, 24h, 48h, and 72h

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China